CLINICAL TRIAL: NCT03458351
Title: Effect of Remote Ischemic Preconditioning on Platelet Activation During Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: RIPC and Platelet Activation on Platelet Activation During Cardiopulmonary Bypass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RIPC_platelet activation
Record Dates: First submitted 2018-02-22; First posted 2018-03-08 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Platelet Dysfunction
Keywords: platelet activation; remote ischemic preconditioning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic preconditioning (Active Comparator): Remote ischemic conditioning after anesthesia induction
  - four cycles of 5 min of ischemia followed by 5 min of reperfusion by inflation to 200 mm Hg and deflation of a blood pressure cuff on the upper arm
  Interventions: Device: Remote ischemic preconditioning
- Sham control (Sham Comparator): The same blood pressure cuff is placed around the upper arm, but the cuff is inflated to 10mm Hg.
  Interventions: Device: Sham control

INTERVENTIONS:
Device: Remote ischemic preconditioning — Four cycles of 5 min of ischemia, which is induced by a blood pressure cuff in the upper arm inflated to 200 mmHg, followed by 5 min of reperfusion, during which the cuff is deflated.
  Arms: Remote ischemic preconditioning
Device: Sham control — The same blood pressure cuff is placed around the upper arm, but the cuff is inflated to 10 mm Hg and ischemic preconditioning is not induced.
  Arms: Sham control

SUMMARY:
In this study, the investigators are going to investigate the effects of remote ischemic preconditioning on platelet activation in patients undergoing cardiac surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
Previous studies reported that remote ischemic conditioning reduce platelet activation in patients with coronary artery disease or patients undergoing ablation for atrial fibrillation. Cardiac surgery with cardiopulmonary bypass has been associated with platelet activation. In this randomized study, investigators are going to compare the effects of remote ischemic preconditioning (RIPC) on platelet activation using flow cytometry in patients undergoing cardiac surgery with cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Preoperative left ventricle ejection fraction < 30%, mechanical ventricular support
* Peripheral vascular disease
* Poorly controlled diabetes mellitus
* NSAIDs within 3 days
* iv heparin within 6 h
* low molecular weight heparin within 24 h
* platelet inhibitor within 24 h
* known thrombocytopenia
* End stage renal disease / hemodialysis
* Active infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Platelet activation measured by CD62P expression using flow cytometry | During 3hour after cardiopulmonary bypass initiation
  CD62P AUC (area under the curve)

SECONDARY OUTCOMES:
Platelet activation measured by CD63 expression using flow cytometry | During 3hour after cardiopulmonary bypass initiation
  CD63 AUC (area under the curve)
Platelet activation measured by monocyte-platelet aggregates (MPA) expression using flow cytometry | During 3hour after cardiopulmonary bypass initiation
  MPA AUC (area under the curve)
Platelet activation measured by PAC1 expression using flow cytometry | During 3hour after cardiopulmonary bypass initiation
  PAC1 AUC (area under the curve)
Platelet activation measured by platelet microparticles (PMP) expression using flow cytometry | During 3hour after cardiopulmonary bypass initiation
  PMP AUC (area under the curve)
ADPtest by Multiplate® platelet function analyser | 3hour after cardiopulmonary bypass initiation
  ADPtest AU
ASPItest by Multiplate® platelet function analyser | 3hour after cardiopulmonary bypass initiation
  ASPItest AU
COLtest by Multiplate® platelet function analyser | 3hour after cardiopulmonary bypass initiation
  COLtest AU

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea